CLINICAL TRIAL: NCT02206802
Title: Minoxidil Response Testing in Females With Female Pattern Hair Loss
Status: Completed | Type: Observational
Sponsor: Applied Biology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AB-IVD-MINOXIDIL-004
Record Dates: First submitted 2014-07-31; First posted 2014-08-01 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Alopecia; Female Pattern Hair Loss
Keywords: Alopecia; Androgenetic Alopecia; Female Pattern Hair Loss; Hair Loss; Minoxidil; Hair Thinning
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plucked hair follicles with visible bulbs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Predicted as non-responders: Patients that the minoxidil response in-vitro diagnostic kit predicted as non-responders. 5% minoxidil topical foam will be administered to subjects in this group.
  Interventions: Drug: 5% minoxidil topical foam
- Predicted as responders: Patients that the minoxidil response in-vitro diagnostic kit predicted as responders. 5% minoxidil topical foam will be administered to subjects in this group.
  Interventions: Drug: 5% minoxidil topical foam

INTERVENTIONS:
Drug: 5% minoxidil topical foam — 5% minoxidil topical foam
  Other Names: Rogaine 5% minoxidil foam; Regaine 5% minoxidil foam

SUMMARY:
The primary purpose of this study is to evaluate the clinical validity of the minoxidil response in-vitro diagnostic kit.

DETAILED DESCRIPTION:
Topical minoxidil is the only US FDA approved drug used for the treatment of AGA in females. While topical minoxidil exhibits a good safety profile, the efficacy in the overall population remains relatively low i.e., 30-40% re-grow hair. To observe significant improvement in hair growth, minoxidil is typically used once daily for a period of at least 24 weeks. Due to the significant time commitment and low response rate, a diagnostic test to identify non-responders prior to initiating therapy would be advantageous.

Minoxidil is converted in the scalp to its active form, minoxidil sulfate, by the sulfotransferase enzyme SULT1A1. The enzyme expression is variable among individuals. We have demonstrated in two prior feasibility studies that the SULT1A1 enzyme activity in plucked hair follicles correlates with minoxidil response in the treatment of AGA and thus can server as a predictive biomarker.

Consequently, we developed a minoxidil response in-vitro diagnostic kit intended to identify non-responders prior to initiating therapy with 5% topical minoxidil foam.

ELIGIBILITY:
Inclusion Criteria:

* Females in overall good health
* Age: 18 or older
* Female pattern hair loss
* Willing to have a mini dot tattoo placed in the target area of the scalp
* Willing to maintain the same hair style, color, shampoo and hair products use, and approximate hair length throughout the study
* Able to give informed consent
* Able to comply with the study requirements for 24 consecutive weeks
* Willing to use an adequate method of birth control (if applicable)
* Negative urine pregnancy test

Exclusion Criteria:

* Previous adverse event from topical minoxidil treatment
* History of hypotension
* Uncontrolled hypertension
* Pregnant, nursing, or planning a pregnancy during the study
* Prior hair transplant
* Uses wigs or hair weaves
* Have used minoxidil (topical or oral) anytime during the past 6 months
* Chronic scalp disorders that require medications
* Uses medication known to cause hair thinning such as Coumadin and anti-depressants/anti-psychotics
* Folliculitis
* Scalp psoriasis
* Seborrheic dermatitis
* Inflammatory scalp conditions such as lichen planopilaris
* Enrolled in any other medical study or has been enrolled in any medical study in the past 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females with Female Pattern Hair Loss - Androgenetic Alopecia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-07; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the minoxidil response in-vitro diagnostic kit to predict at baseline the change in Target Area Hair Count | baseline to week 24
  Number of hairs measured in the target area by macrophotography.
Sensitivity and specificity of the minoxidil response in-vitro diagnostic kit to predict at baseline the subjects ratings | baseline to week 24

SECONDARY OUTCOMES:
Sensitivity and specificity of the minoxidil response in-vitro diagnostic kit to predict at baseline the change in Target Area Hair Count | baseline to week 12
  Number of hairs measured in the target area by macrophotography.
Sensitivity and specificity of the minoxidil response in-vitro diagnostic kit to predict at baseline the treatment efficacy evaluated by expert panel review of global photographs assessing hair regrowth | baseline to week 24
Sensitivity and specificity of the minoxidil response in-vitro diagnostic kit to predict at baseline the mean change in non-vellus hair diameter in the target region | baseline to week 24
Mean change in minoxidil sulfotransferase activity in plucked hairs as measured by the minoxidil response in-vitro diagnostic kit | baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Keene, MD, Principal Investigator — Physicians Hair Institute; Flavio Grasso, MD, Principal Investigator — Istituto Medico Tricologico/Studi Life Cronos; Rodney Sinclair, MD, Principal Investigator — Sinclair Dermatology; Rachita Dhurat, MD, Principal Investigator — LTM Medical College & Hospital
Locations (5):
- United States (2):
  - Physicians Hair Institute, Tucson, Arizona
  - Tennessee Clinical Research Center, Nashville, Tennessee
- Sinclair Dermatology, East Melbourne, Australia
- LTM Medical College & Hospital, Mumbai, India
- Istituto Medico Tricologico/Studi Life Cronos, Florence, Italy

REFERENCES:
- [Background] Roberts J, Desai N, McCoy J, Goren A. Sulfotransferase activity in plucked hair follicles predicts response to topical minoxidil in the treatment of female androgenetic alopecia. Dermatol Ther. 2014 Jul-Aug;27(4):252-4. doi: 10.1111/dth.12130. Epub 2014 Apr 28. PMID 24773771
- [Background] Goren A, Castano JA, McCoy J, Bermudez F, Lotti T. Novel enzymatic assay predicts minoxidil response in the treatment of androgenetic alopecia. Dermatol Ther. 2014 May-Jun;27(3):171-3. doi: 10.1111/dth.12111. Epub 2013 Nov 27. PMID 24283387
- [Background] Buhl AE, Waldon DJ, Baker CA, Johnson GA. Minoxidil sulfate is the active metabolite that stimulates hair follicles. J Invest Dermatol. 1990 Nov;95(5):553-7. doi: 10.1111/1523-1747.ep12504905. PMID 2230218
- [Background] Messenger AG, Rundegren J. Minoxidil: mechanisms of action on hair growth. Br J Dermatol. 2004 Feb;150(2):186-94. doi: 10.1111/j.1365-2133.2004.05785.x. PMID 14996087